CLINICAL TRIAL: NCT00051389
Title: ACE Inhibition and Novel Cardiovascular Risk Factors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 155; R01HL068901 (NIH)
Record Dates: First submitted 2003-01-09; First posted 2003-01-13 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2008-01

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension | interventions — Fosinopril

INTERVENTIONS:
Drug: Fosinopril

SUMMARY:
To determine the effects of an angiotensin converting enzyme inhibitor (ACE inhibitor), fosinopril, on multiple blood markers in 286 adults at high risk for cardiovascular disease.

DETAILED DESCRIPTION:
BACKGROUND:

Angiotensin converting enzyme inhibitors (ACE inhibitors) may prevent cardiovascular events in high risk persons and improve skeletal muscle function in heart failure patients by means of mechanisms that are independent of blood pressure changes. However, there is limited knowledge of all the mechanisms underlying the therapeutic benefits of ACE inhibition. ACE inhibitors may favorably modify markers of fibrinolysis, inflammation, endothelial function, and extracellular tissue remodeling, all of which are associated with atherosclerosis and cardiovascular disease. But, clinical trial evidence on these effects is limited. In addition, polymorphisms of the ACE, angiotensinogen, PAI-1 and IL-6 genes may modify the therapeutic response to ACE inhibitors.

DESIGN NARRATIVE:

This was a double-blind cross-over, randomized, placebo controlled trial in 286 persons with high cardiovascular risk to compare the effects of 6 months of treatment with fosinopril and 6 months with placebo on the following primary outcomes: plasma plasminogen activator inhibitor-1 (PAI-1) antigen, C- reactive protein (CRP), interleukin-6 (IL-6) and soluble vascular cell adhesion molecule-1 (sVCAM-1). The secondary objectives were (a) to assess the effects of fosinopril on IL-6/IL-6 Soluble Receptor ratio, PAI-1 activity, tissue plasminogen activator (TPA) antigen, fibrinogen, endothelin-1, TNF-alpha, soluble intercellular cell adhesion molecule-1 (sICAM-1), E-selectin, matrix metalloproteinase-1 (MMP-1) and tissue inhibitor of metalloproteinase-1 (TIMP-1); and (b) to explore the effects of ACE, angiotensinogen, PAI-1, and IL-6 gene polymorphisms on these biomarkers, and test the interaction of the gene polymorphisms with the effects of fosinopril. The study had sufficient power to detect small changes in several biomarkers compared to placebo. The assessment of these biological mechanisms had clinical relevance for identifying the patients who may benefit the most from ACE inhibition. While the focus of the study was on novel cardiovascular risk factors, the results may also have future implications for developing new indications for ACE inhibitors, such as, for example, the prevention of age-related muscle wasting and physical disabilities in older persons, for which inflammation may be a causal factor.

ELIGIBILITY:
No eligibility criteria

Ages: 55 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-02; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marco Pahor — Wake Forest University Health Sciences

REFERENCES:
- [Background] Cesari M, Kritchevsky SB, Baumgartner RN, Atkinson HH, Penninx BW, Lenchik L, Palla SL, Ambrosius WT, Tracy RP, Pahor M. Sarcopenia, obesity, and inflammation--results from the Trial of Angiotensin Converting Enzyme Inhibition and Novel Cardiovascular Risk Factors study. Am J Clin Nutr. 2005 Aug;82(2):428-34. doi: 10.1093/ajcn.82.2.428. PMID 16087989